CLINICAL TRIAL: NCT01808872
Title: Clinical Sensitivity and Specificity Study of AQT90 FLEX BNP and NT-proBNP
Brief Title: Clinical Performance Evaluation of AQT90 FLEX BNP and NT-proBNP
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-043652
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples are retained only for this study (troubleshooting purposes).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure

SUMMARY:
The AQT90 FLEX B-type Natriuretic Peptide (BNP) and N-terminal pro B-type natriuretic peptide (NT-proBNP) Tests are in vitro diagnostic assays intended as an aid in the diagnosis and assessment of the severity of heart failure in point-of-care and laboratory settings. The purpose of the study is to establish the clinical performance of the AQT90 FLEX BNP and NT-proBNP assays for both whole blood and plasma in the intended use population.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 21 years of age or older
* Subject is able to understand information given, and willing and able to voluntarily give their consent to participate in this study
* Subject has diagnosis of heart failure

Exclusion Criteria:

* Subject has Acute Coronary Syndrome (ACS)
* Subject has been diagnosed and/or treated for malignancy within past 6 months
* Subject has had cardiac surgery within the past 4 weeks
* Subject claim of pregnancy
* Subject's prior participation in this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 21 years of age or older with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Determination of the clinical sensitivity and specificity of the AQT90 FLEX BNP and NT-proBNP assays at the clinical cut-off in heart failure patients | Single blood draw upon study entry
  Clinical sensitivity and specificity with 95 % confidence intervals of the AQT90 FLEX BNP and NT-proBNP assays will be determined at the clinical cut-off in heart failure patients divided by age, gender and New York Heart Association (NYHA) functional classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States